CLINICAL TRIAL: NCT06101329
Title: A Phase 2, Open-label, Multicenter, Randomized Study to Evaluate the Pharmacokinetics, Safety, and Acceptability of Twice Yearly Long-acting Subcutaneous Lenacapavir for Pre-Exposure Prophylaxis in Cisgender Women in the United States
Brief Title: Study of Lenacapavir and Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) in Prevention of HIV in Cisgender Women in the United States (HPTN 102)
Acronym: PURPOSE 3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GS-US-528-6020
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pre-Exposure Prophylaxis of HIV Infection
MeSH Terms: interventions — lenacapavir; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized Phase: Lenacapavir (LEN) Group (Experimental): Participants will receive subcutaneous (SC) lenacapavir (LEN) 927 mg on Day 1 and Week 26 and oral LEN 600 mg on Days 1 and 2.
  Interventions: Drug: Lenacapavir Tablet; Drug: Lenacapavir Injection
- Randomized Phase: Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) Group (Experimental): Participants will receive oral F/TDF (200/300 mg) daily for 52 weeks.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF)
- PK Tail Phase: F/TDF (Experimental): After the completion of the Randomized Phase, participants in LEN group will be transitioned to receive F/TDF and participants in F/TDF group will continue to receive F/TDF in the PK Tail Phase. All participants will receive F/TDF, once daily for 78 weeks beginning 26 weeks after the last LEN injection.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF)

INTERVENTIONS:
Drug: Lenacapavir Tablet — Tablets administered orally without regard of food
  Other Names: GS-6207
  Arms: Randomized Phase: Lenacapavir (LEN) Group
Drug: Lenacapavir Injection — Injection administered subcutaneously
  Other Names: GS-6207; Yeztugo®
  Arms: Randomized Phase: Lenacapavir (LEN) Group
Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) — 200/300mg fixed dose combination (FDC) tablets administered orally
  Other Names: Truvada®
  Arms: PK Tail Phase: F/TDF; Randomized Phase: Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) Group

SUMMARY:
The goal of this clinical study is to look at how lenacapavir (LEN) passes through the body and to assess the safety of LEN and emtricitabine/tenofovir disoproxil fumarate (F/TDF) for prevention of HIV in the cisgender women in the US.

The primary objectives of this study are: 1) to characterize the pharmacokinetics (PK) of LEN in United States (US) cisgender women; 2) to evaluate the safety of LEN and F/TDF for pre-exposure prophylaxis (PrEP) in US cisgender women; and 3) to evaluate the general acceptability of LEN injections and oral F/TDF in US cisgender women.

ELIGIBILITY:
Key Inclusion Criteria:

* Report at least 1 episode of condomless vaginal or anal sex with a cisgender man in the 12 months before enrollment.
* Hepatitis B virus (HBV) surface antigen (HBsAg) negative.
* Self-report one or more of the following in the past 12 months (except for incarceration, which could have occurred in the past 5 years):

  1) Noninjection recreational drug use (ecstasy, cocaine, crack cocaine, methamphetamine, ketamine, 3,4-methylenedioxy-methamphetamine, or prescription drugs apart from those prescribed by a licensed provider); 2) Alcohol dependence (defined as Cut Down, Annoyed, Guilty, and Eye Opener score of 2); binge-drinking, defined as 4 or more drinks at a time; 3) History of STIs, such as gonorrhea, chlamydia, or syphilis; 4) Exchange of sex for commodities, such as drugs, money, or shelter; 5) Incarceration (jail or prison > 24 hours within the past 5 years); 6) Two or more sexual partners who were assigned male at birth; 7) Sexual partner assigned male at birth with history of either injection or noninjection recreational drug use, sexually transmitted infections (STIs), human immunodeficiency virus (HIV) diagnosis or unknown HIV status, additional sex partners during the course of his sexual relationship with the individual, or incarceration (jail or prison > 24 hours within the past 5 years)
* Negative local rapid HIV-1/2 antibody (Ab)/antigen (Ag) test, central HIV-1/2 Ab/Ag, and HIV-1 RNA quantitative nucleic acid amplification testing (NAAT).
* Estimated glomerular filtration rate (GFR) at least 60 mL/min at screening according to the Cockcroft-Gault formula for creatinine clearance (CLcr).

Key Exclusion Criteria:

* Self-reported history of previous positive results on an HIV test.
* One or more reactive or positive HIV test result at screening or enrollment, even if HIV infection is not confirmed.
* Past or current participation in HIV vaccine or HIV broadly neutralizing antibody study unless individual provides documentation of receipt of placebo (ie, not active product).
* Prior use of long-acting systemic pre-exposure prophylaxis (PrEP) (including cabotegravir (CAB) or islatravir studies).
* Acute viral hepatitis A or acute or chronic hepatitis B or C infection.
* Severe hepatic impairment or a history of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, variceal bleeding, etc).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender female
Enrollment: 253 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Ctrough for Lenacapavir (LEN) at the End of Week 26 | Week 26
  Ctrough is defined as the concentration at the end of the dosing interval.
PK Parameter: Ctrough for LEN at the End of Week 52 | Week 52
  Ctrough is defined as the concentration at the end of the dosing interval.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 30 days post last dose at Week 78
Percentage of Participants Experiencing Treatment-emergent Clinical Laboratory Abnormalities | First dose date up to 30 days post last dose at Week 78
General Acceptability of LEN and F/TDF as PrEP as Assessed by Percentage of Participants with Acceptability Questionnaire Responses | Up to Week 52
  To assess the acceptability of the study drug, participants will complete the questionnaire including a question on general acceptability of the assigned study drug on an ordinal 5-category scale with a response of: Completely unacceptable, Unacceptable, No opinion, Acceptable, or Completely acceptable.
Satisfaction With Use of LEN and F/TDF as PrEP as Assessed by Percentage of Participants with Satisfaction Questionnaire Responses | Up to Week 52
  To assess the satisfaction with use of the study drug, participants will complete the questionnaire including a question on satisfaction with use of the assigned study drug on an ordinal 5-category scale with a response of: Very satisfied, Satisfied, Neutral, Dissatisfied, or Very dissatisfied.
Willingness to Use LEN and F/TDF as PrEP as Assessed by Percentage of Participants with Willingness to Use Questionnaire Responses | Up to Week 52
  To assess the willingness to use the study drug, participants will complete the questionnaire including a question on willingness to use the assigned study drug on an ordinal 5-category scale with a response of: Definitely Yes, Probably yes, Not sure/undecided, Probably No, or Definitely No.

SECONDARY OUTCOMES:
Number of Participants with Adherence to LEN, as Assessed by on-time LEN Injections Received | Up to Week 26
Number of Participants with Adherence to F/TDF, as Assessed by Adherence Levels Based on Tenofovir diphosphate (TFV-DP) Concentrations in Dried Blood Spot (DBS) | Up to Week 78

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (11):
- United States (11):
  - UAB, 1917 Research Clinic, Birmingham, Alabama
  - UCSD Antiviral Research Center (AVRC), San Diego, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Ponce de Leon Center Clinical Research Site, Atlanta, Georgia
  - Fenway Health, Boston, Massachusetts
  - Rutgers New Jesey Medical School - Clinical Research Center, Newark, New Jersey
  - Cornell Clinical Trials Unit, New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York
  - Harlem Prevention Center CRS, New York, New York
  - ICAP at Columbia University - Bronx Prevention Center, The Bronx, New York
  - NC TraCS Institute - CTRC; University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Penn Prevention Research Unit, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06101329